CLINICAL TRIAL: NCT02675478
Title: A Phase 1, Open-Label, Dose Escalation Study of Quizartinib, An Oral FLT3 Inhibitor, in Japanese Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Phase 1 Study of Quizartinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC220-A-J101
Record Dates: First submitted 2016-02-02; First posted 2016-02-05 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2018-11

CONDITIONS: Relapsed AML; Refractory AML
Keywords: AML; phase 1; oncology
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AC220 (Experimental): This study will follow a mCRM (modified continual reassessment method) + EWOC (Escalation with Overdose Control) design.
  Interventions: Drug: AC220

INTERVENTIONS:
Drug: AC220

SUMMARY:
This is a dose escalation study to evaluate the safety, tolerability, and pharmacokinetics of quizartinib for Japanese acute myeloid leukemia (AML) subjects.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory AML
* AML for which no standard treatment is available
* ECOG Performance Status (PS) of 0 to 2

Exclusion Criteria:

* Acute Promyelocytic Leukemia
* chronic myelogenous leukemia in blast phase (BCR-ABL fusion gene positive)
* History of other malignancies within 3 years prior to enrollment, except curatively treated in-situ carcinoma, AML, or MDS.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-02; Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
number of subjects experiencing adverse events | first dose to follow-up, approximately 1 year
Cmax of quizartinib and its active metabolite | Cycle 1: Days 1, 2, 4, 8, 11, 15, 16, 18, 22, 28; Cycle 2 and on: Days 1, 15
  Evaluate the pharmacokinetics of quizartinib and its active metabolite, AC886 by Cmax, Tmax, AUCtau, Cmax,ss, Ctrough, Tmax,ss, AUCtau,ss.
Tmax of quizartinib and its active metabolite | Cycle 1: Days 1, 2, 4, 8, 11, 15, 16, 18, 22, 28; Cycle 2 and on: Days 1, 15
  Evaluate the pharmacokinetics of quizartinib and its active metabolite, AC886 by Cmax, Tmax, AUCtau, Cmax,ss, Ctrough, Tmax,ss, AUCtau,ss.
AUCtau of quizartinib and its active metabolite | Cycle 1: Days 1, 2, 4, 8, 11, 15, 16, 18, 22, 28; Cycle 2 and on: Days 1, 15
  Evaluate the pharmacokinetics of quizartinib and its active metabolite, AC886 by Cmax, Tmax, AUCtau, Cmax,ss, Ctrough, Tmax,ss, AUCtau,ss.
Cmax,ss of quizartinib and its active metabolite | Cycle 1: Days 1, 2, 4, 8, 11, 15, 16, 18, 22, 28; Cycle 2 and on: Days 1, 15
  Evaluate the pharmacokinetics of quizartinib and its active metabolite, AC886 by Cmax, Tmax, AUCtau, Cmax,ss, Ctrough, Tmax,ss, AUCtau,ss.
Ctrough of quizartinib and its active metabolite | Cycle 1: Days 1, 2, 4, 8, 11, 15, 16, 18, 22, 28; Cycle 2 and on: Days 1, 15
  Evaluate the pharmacokinetics of quizartinib and its active metabolite, AC886 by Cmax, Tmax, AUCtau, Cmax,ss, Ctrough, Tmax,ss, AUCtau,ss.
Tmax,ss of quizartinib and its active metabolite | Cycle 1: Days 1, 2, 4, 8, 11, 15, 16, 18, 22, 28; Cycle 2 and on: Days 1, 15
  Evaluate the pharmacokinetics of quizartinib and its active metabolite, AC886 by Cmax, Tmax, AUCtau, Cmax,ss, Ctrough, Tmax,ss, AUCtau,ss.
AUCtau,ss of quizartinib and its active metabolite | Cycle 1: Days 1, 2, 4, 8, 11, 15, 16, 18, 22, 28; Cycle 2 and on: Days 1, 15
  Evaluate the pharmacokinetics of quizartinib and its active metabolite, AC886 by Cmax, Tmax, AUCtau, Cmax,ss, Ctrough, Tmax,ss, AUCtau,ss.

SECONDARY OUTCOMES:
FMS-like tyrosine kinase-3 / internal tandem duplication FLT3/ITD allelic ratio | Cycle 1: Days 1, 2, 8, 15
  Exploratory assessment of quizartinib-related biomarkers such as FLT3-ITD allelic ratio, PIA assessment.
PIA assessment | Cycle 1: Days 1, 2, 8, 15
  Exploratory assessment of quizartinib-related biomarkers such as FLT3-ITD allelic ratio, PIA assessment.
bone marrow findings | Cycle 1: Days 15, 28; Cycle 2 and on: Day 28
  Exploratory analyses of tumor response to quizartinib based on bone marrow findings, absolute neutrophil count, and platelet count.
absolute neutrophil count | Cycle 1: Days 15, 28; Cycle 2 and on: Day 28
  Exploratory analyses of tumor response to quizartinib based on bone marrow findings, absolute neutrophil count, and platelet count.
platelet count | Cycle 1: Days 15, 28; Cycle 2 and on: Day 28
  Exploratory analyses of tumor response to quizartinib based on bone marrow findings, absolute neutrophil count, and platelet count.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Usuki K, Handa H, Choi I, Yamauchi T, Iida H, Hata T, Ohwada S, Okudaira N, Nakamura K, Sakajiri S. Safety and pharmacokinetics of quizartinib in Japanese patients with relapsed or refractory acute myeloid leukemia in a phase 1 study. Int J Hematol. 2019 Dec;110(6):654-664. doi: 10.1007/s12185-019-02709-8. Epub 2019 Jul 29. PMID 31359361